CLINICAL TRIAL: NCT05398393
Title: An Experimental Study on the Effect of Tenofovir Amibufenamide on Blood Lipid During Anti-HBV Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Jin Ye, professor, chief doctor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHCT21612
Record Dates: First submitted 2022-03-10; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Hepatitis B, Chronic; Lipid Disorder
Keywords: Tenofovir Amibufenamide
MeSH Terms: conditions — Hepatitis B, Chronic; Lipid Metabolism Disorders | interventions — Amlodipine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Other): normal blood lipid level at baseline
  Interventions: Drug: oral Tenofovir Amibufenamide 25mg each day
- group B1 (Other): baseline blood lipid is elevated and treat with lipid-lowering drugs
  Interventions: Drug: oral Tenofovir Amibufenamide 25mg each day; Drug: lipid lowering drugs (e.g. Atorvastatin and amlodipine.)
- group B2 (Other): baseline blood lipid is elevated and without lipid-lowering drugs treatment
  Interventions: Drug: oral Tenofovir Amibufenamide 25mg each day

INTERVENTIONS:
Drug: oral Tenofovir Amibufenamide 25mg each day — patients in three groups respectively take one tablet of Tenofovir Amibufenamide(25mg) every day
Drug: lipid lowering drugs (e.g. Atorvastatin and amlodipine.) — lipid lowering drugs, , patients in group B1 continue take lipid lowering drugs
  Arms: group B1

SUMMARY:
In June 2021, Chinese Food and Drug Administration approved the launch of the self-developed new drug Tenofovir Amibufenamide(TMF). TMF is a new second generation of tenofovir(TFV) and its effect on blood lipids is unclear. Our study aims to figure out the effect of TMF on serum lipid level in the process of antiviral therapy for chronic hepatitis B patients.

DETAILED DESCRIPTION:
In June 2021, Chinese Food and Drug Administration approved the launch of the self-developed new drug Tenofovir Amibufenamide(TMF). TMF is the phosphoramidite precursor of Tenofovir, belonging to the nucleoside reverse transcriptase and owning higher cell membrane penetration rate, which make it easier to enter hepatocytes and achieve liver-targeted therapy. Meanwhile, TMF can effectively improve drug stability in plasma and reduce systemic tenofovir(TFV) exposure, and make long-term treatment safer.

Previous studies have shown that tenofovir disoproxil (TDF), the first generation of TFV, had the effect of lowering blood lipids. While patients who switched to tenofovir alafenamide (TAF), the second generation of TFV, had elevated blood lipids. TMF is a new second generation of TFV and its effect on blood lipids is unclear. Our study aims to figure out the effect of TMF on serum lipid level in the process of antiviral therapy for chronic hepatitis B patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old;
2. Chronic hepatitis B patients who meet the CHB diagnostic criteria of "Guidelines for the Prevention and Treatment of Chronic Hepatitis B (Chinese 2019 version)";
3. HBV-DNA can be detected (≥20IU/mL);
4. With or without liver cirrhosis caused by hepatitis B;
5. The treatment plan is TMF antiviral therapy, and no other antiviral drugs are used for at least 1 year before;
6. The clinical data are relatively complete, and the follow-up time reaches 24 weeks (6 months).

Exclusion Criteria:

1. Patients with primary liver cancer or liver metastases;
2. Combined with hepatitis A virus, hepatitis C virus, hepatitis D virus, hepatitis E virus and human immunodeficiency virus infection;
3. Combined with alcoholic liver disease, drug-induced liver disease, autoimmune liver disease and liver disease caused by other factors;
4. History of treatment of dysglycemia and dyslipidemia;
5. Patients with lactose intolerance;
6. Pregnant women and lactating women;
7. Patients with other serious systemic diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
change from baseline HBV-DNA at 1/3/6/12month | baseline, follow up of 1,3,6,12month
  test virological response rate
change from baseline level of blood lipid at 1/3/6/12month | baseline, follow up of 1,3,6,12month
  test blood lipid level

SECONDARY OUTCOMES:
change from baseline serum calcium at 6/12month | baseline, follow up of 6,12month
  test blood serum calcium
change from baseline serum phosphorus at 6/12month | baseline, follow up of 6,12month
  test blood serum phosphorus

OTHER OUTCOMES:
change from baseline liver stiffness measurement at 6/12month | baseline, follow up of 6,12month
  test liver stiffness measurement and controlled attenuation parament through transient elastography(FibroTouch)
ultrasonography | baseline, follow up of 6,12month
  liver ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Wuhan Union hosipital, Principal Investigator — Affiliated to Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Wuhan Union hosipital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared including study protocol, statistical analysis, informed consent plan, clinical study report and analytic code
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: the data will be available after June 2023
Access Criteria: academic exchange
URL: http://www.whuh.com/

REFERENCES:
- [Result] Suzuki K, Suda G, Yamamoto Y, Furuya K, Baba M, Nakamura A, Miyoshi H, Kimura M, Maehara O, Yamada R, Kitagataya T, Yamamoto K, Shigesawa T, Nakamura A, Ohara M, Kawagishi N, Nakai M, Sho T, Natsuizaka M, Morikawa K, Ogawa K, Ohnishi S, Sakamoto N; NORTE Study Group. Tenofovir-disoproxil-fumarate modulates lipid metabolism via hepatic CD36/PPAR-alpha activation in hepatitis B virus infection. J Gastroenterol. 2021 Feb;56(2):168-180. doi: 10.1007/s00535-020-01750-3. Epub 2020 Nov 19. PMID 33211179
- [Result] Lacey A, Savinelli S, Barco EA, Macken A, Cotter AG, Sheehan G, Lambert JS, Muldoon E, Feeney E, Mallon PW, Tinago W; UCD ID Cohort Study. Investigating the effect of antiretroviral switch to tenofovir alafenamide on lipid profiles in people living with HIV. AIDS. 2020 Jul 1;34(8):1161-1170. doi: 10.1097/QAD.0000000000002541. PMID 32310899
- [Result] Ikeda M, Wakabayashi Y, Okamoto K, Yanagimoto S, Okugawa S, Moriya K. Changing trends in lipid profile and biomarkers of renal function and bone metabolism before and after switching from tenofovir disoproxil fumarate to tenofovir alafenamide: a prospective observational study. AIDS Res Ther. 2021 May 27;18(1):30. doi: 10.1186/s12981-021-00354-y. PMID 34044856
- [Result] Li M, Zhou L, Dorsey HG, Musoff C, Jnr DA, Schoen N, Djan K, Paintsil E. Tenofovir alafenamide does not inhibit mitochondrial function and cholesterol biosynthesis in human T lymphoblastoid cell line. Antiviral Res. 2020 Nov;183:104948. doi: 10.1016/j.antiviral.2020.104948. Epub 2020 Sep 24. PMID 32980447

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT05398393/Prot_SAP_ICF_000.pdf